CLINICAL TRIAL: NCT00421096
Title: Stage IB2 to IVA Uterine Cervical Cancer: Phase 2 Study to Assess a New Therapeutic Sequence Associating a Radiochemotherapy Followed by Adjuvant Chemotherapy Based on Gemcitabine
Brief Title: Radiochemotherapy Followed by Adjuvant Chemotherapy Based on Gemcitabine in Uterine Cervical Cancer
Acronym: GEMCOL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Problems of recruitment
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCOL 0401
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Uterine Cervical Cancer
Keywords: uterine cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Gemcitabine; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient with cervix cancer (Experimental): will receive gemcitabine + cisplatin + radiotherapy
  Interventions: Drug: Gemcitabine; Procedure: Radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — 125 mg/m² at day 1, 8, 15, 21 and 28, 2 hours before radiotherapy.
Procedure: Radiotherapy — 45Gy (5 x 1,8Gy/week) on pelvic area +/- boost (10 to 15Gy)
  +/- 45Gy (5 x 1,8Gy/week)on lumbo-aortic area
Drug: Cisplatin — 40 mg/m² at day 1, 8, 15, 21 and J28 before Gemcitabine and with a hyperhydration

SUMMARY:
The scope of the trial is to assess the efficacy of the association gemcitabine-cisplatin + radiotherapy followed by an adjuvant chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Cervical uterine cancer (epidermoid or adenocarcinoma, stage:from IB> or = 4 cm to IV, according to FIGO classification) histologically proven
* Measurable lesions,clinically and by MRI assessed
* PS-WHO < or = 2 ou Karnofsky Index >70 per cent
* Life expectancy > 3 months
* Hematologic function: leukocytes < or = 3 G/l, polynuclear neutrophil leukocytes > or = 1.5 G/l, platelets > or = 100 G/l, hemoglobin > or = 10 g/dl
* Hepatic function: ASAT and ALAT < 2.5 ULN
* Renal function: creatininemia < 1.5 ULN, clearance > 60 ml/min
* No prior chemotherapy or radiotherapy
* Contraception
* Written informed consent signed

Exclusion Criteria:

* Stage IB < 4 cm or IVB
* Other histology than epidermoid or adenocarcinoma
* Distant metastases, including sus-clavicular adenopathy
* Contraindication to MRI
* Pregnant or lactating woman
* Auto-immune disease
* Peripheric neuropathy, autograft or homograft, psychiatric disease
* Prior cancer (except cutaneous basocellular carcinoma and uterine cervical carcinoma in situ)
* Active infection
* Other clinical trial with an experimental drug
* Known positive serology (HIV, HbC, HbS)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 3 years after the end of study treament

SECONDARY OUTCOMES:
Global survival | 5 years after the end of study treatment
safety | untill 5 years after study treatment

CONTACTS AND LOCATIONS:
Overall Officials: BELKACEMI Yazid, MD, Principal Investigator — Centre Oscar Lambret
Locations (2):
- France (2):
  - Centre Leonard de Vinci, Dechy
  - Centre Oscar Lambret, Lille